CLINICAL TRIAL: NCT04726085
Title: Efficacy of Ibuprofen Versus Indomethacin as Perioperative Prophylactic Treatment Following Emergent Cerclage Placement for Pregnancy Prolongation: A Randomized Controlled Trial
Brief Title: Ibuprofen Versus Indomethacin Following Emergent Cerclage Placement
Acronym: TOCO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigative team moved institutions
Sponsor: Woman's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RP-20-028
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Preterm Labor
Keywords: cerclage
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Indomethacin; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ibuprofen (Active Comparator): Ibuprofen 600 mg q6 hours for 24 hours- total dose of 2400mg- after emergent cerclage placement
  Interventions: Drug: Ibuprofen 2400mg
- Indomethacin (Active Comparator): Indomethacin 50 mg q8 hours for 24 hours- total dose of 150mg- after emergent cerclage placement
  Interventions: Drug: Indomethacin 150mg

INTERVENTIONS:
Drug: Indomethacin 150mg — Patients will be randomized to either received perioperative indomethacin or ibuprofen at the time of their emergent cerclage placement for 24 hours following surgery. Patient will be followed up through our electronic medical record system to determine gestational latency to evaluate if ibuprofen is inferior to indomethacin.
  Arms: Indomethacin
Drug: Ibuprofen 2400mg — Patients will be randomized to either received perioperative indomethacin or ibuprofen at the time of their emergent cerclage placement for 24 hours following surgery. Patient will be followed up through our electronic medical record system to determine gestational latency to evaluate if ibuprofen is inferior to indomethacin.
  Arms: Ibuprofen

SUMMARY:
Cervical insufficiency is defined as painless cervical dilation in the second trimester. Cervical insufficiency can ultimately lead to second trimester loss of pregnancy. Cerclages are utilized in pregnancies affected by cervical insufficiency in order to prolong gestational latency. There have been several studies investigating the efficacy of perioperative medications for cerclage placement and the effects they have on gestational latency. Some such studies have found that perioperative indomethacin in combination with antibiotics have significantly increased gestational latency when compared to placebo. Indomethacin has traditionally been the tocolytic of choice with cerclage placement. At our hospital, ibuprofen has been the tocolytic of choice for cerclage placement secondary to pharmacy availability. Our study aims to evaluate whether gestational latency differs among patients undergoing emergent cerclage whether they receive perioperative ibuprofen or indomethacin.

ELIGIBILITY:
Inclusion Criteria:

* Viable, singleton pregnancy
* ≥ 18 years old
* Gestational age 16 weeks 0/7 days - 23 week 6/7 days (inclusive)
* Intact membranes at time of enrollment
* Planning to deliver at Woman's Hospital
* Exam or ultrasound indicated cerclage placement

Exclusion Criteria:

* Contraindication to treatments (i.e. ibuprofen or indomethacin)
* Unwilling to be randomized to treatment
* Prophylactic cerclage placement
* Temperature greater than 100.4
* Known major fetal congenital anomaly
* Prior cerclage placement during the current pregnancy
* Recent (within 7 days) receipt of ibuprofen or indomethacin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2023-11-06 (Actual)

PRIMARY OUTCOMES:
Gestational latency | From cerclage placement to delivery
  Days from cerclage placement to delivery, assessed up to 26 weeks

SECONDARY OUTCOMES:
Preterm birth | At delivery
  Birth before 37 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Simmons, DO, Principal Investigator — Woman's Hospital, Louisiana
Locations (1):
- Woman's Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No